CLINICAL TRIAL: NCT06017817
Title: Regular Home-use of Antibacterial Photodynamic Therapy in the Management of Peri-implantitis
Brief Title: Antibacterial Photodynamic Therapy in the Management of Peri-implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nilminie Rathnayake (Industry)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Nilminie Rathnayake, Principal Investigator, Koite Health Oy
Organization: Koite Health Oy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEALTHIER
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Peri-Implantitis; Plaque, Dental
Keywords: Lumoral; Lumorinse; Antibacterial photodynamic therapy (aBPT); aMMP-8; Plaque control
MeSH Terms: conditions — Peri-Implantitis; Dental Plaque | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: 80 subjects in total are recruited to this study: 40 subjects in the non-surgical treatment (NST), of which 20 participants in the NST Study group (NST-1) and 20 participants in the NST Control group (NST-2), and 40 subjects in the surgical treatment (ST), of which 20 participants in the ST Study group (ST-1) and 20 participants in the ST Control group (ST-2).
Who Masked: Participant, Investigator
Masking Description: The first assessments will be made before randomization.
  After the randomization, there is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-surgical treatment, Study group (NST-1) (Experimental): Lumoral Treatment; Standard, non-surgical anti-infective treatment by scaling and root planing (SRP); and Standard oral hygiene instructions for electric toothbrushing, interdental brush, and dental floss use.
  Interventions: Device: Lumoral Treatment; Procedure: Standard oral hygiene instructions; Procedure: Scaling and root planing (SRP
- Non-surgical treatment, Control group (NST-2) (Active Comparator): Standard, non-surgical anti-infective treatment by scaling and root planing (SRP); and Standard oral hygiene instructions for electric toothbrushing, interdental brush, and dental floss use.
  Interventions: Procedure: Standard oral hygiene instructions; Procedure: Scaling and root planing (SRP
- Surgical treatment, Study group (ST-1) (Experimental): Lumoral Treatment; Surgical anti-infective peri-implantitis treatment; and Standard oral hygiene instructions for electric toothbrushing, interdental brush, and dental floss use.
  Interventions: Device: Lumoral Treatment; Procedure: Standard oral hygiene instructions; Procedure: surgical anti-infective peri-implantitis treatment
- Surgical treatment, Control group (ST-2) (Active Comparator): Surgical anti-infective peri-implantitis treatment; and Standard oral hygiene instructions for electric toothbrushing, interdental brush, and dental floss use.
  Interventions: Procedure: Standard oral hygiene instructions; Procedure: surgical anti-infective peri-implantitis treatment

INTERVENTIONS:
Device: Lumoral Treatment — Anti-infective photodynamic therapy for plaque-induced oral conditions
  Arms: Non-surgical treatment, Study group (NST-1); Surgical treatment, Study group (ST-1)
Procedure: Standard oral hygiene instructions — Standard oral hygiene instructions for electric toothbrushing, interdental brush, and dental floss use
Procedure: Scaling and root planing (SRP — non-surgical anti-infective treatment by scaling and root planing
  Arms: Non-surgical treatment, Control group (NST-2); Non-surgical treatment, Study group (NST-1)
Procedure: surgical anti-infective peri-implantitis treatment — surgical anti-infective peri-implantitis treatment
  Arms: Surgical treatment, Control group (ST-2); Surgical treatment, Study group (ST-1)

SUMMARY:
This early-stage study is designed to determine the efficacy of the Lumoral method in periimplantitis. Improved supragingival plaque control can help to also sustain subgingival plaque management in the long term. In addition, the device might have a photobiomodulation effect on periodontal tissues, thus impacting osseointegration.

DETAILED DESCRIPTION:
Clinical signs of inflammation in peri-implantitis include bleeding on probing, suppuration, increased probing depth, and radiographic signs of bone loss. Currently, the best treatment options for peri-implantitis include non-surgical methods of biofilm removal in the supra-mucosal area around implants, and comprehensive guidance on self-performed infection control procedures. With more advanced peri-implantitis, anti-infective surgical treatment protocol would be needed.

Matrix metalloproteinase 8 (MMP-8) has been found to be elevated in association with oral infections, such as periodontitis and peri-implantitis. The level of active MMP-8 (aMMP-8) can detect to determine tissue health and to assess inflammation, and can easily be measured during a regular dental appointment with a chairside test.

The Lumoral Treatment is a CE-marked medical device developed to provide a potent, targeted antibacterial action on dental plaque in a home environment. The method mechanism of action is antibacterial photodynamic therapy (aPDT). The method is used by swishing a mouth rinse, which has a strong adherence to dental plaque. The plaque-adhered photoactive mouth rinse can be activated by a simple-to-use light applicator. Preliminary results have shown a promising anti-inflammatory response in addition to plaque reduction.

ELIGIBILITY:
Inclusion Criteria:

* PPD ≥6 mm and marginal bone loss >3 mm
* Dental implants collected and clinically characterized according to Lähteenmäki et al. CEDR-22
* Agreement to participate in the study and to sign a written consent form
* Able to co-operate with the treatment protocol and avoid any other oral hygiene measures outside of the study protocol

Exclusion Criteria:

* Presence of any physical limitation or restriction that might restrict Lumoral use
* Unwilling to participate in the study
* Pregnancy or lactation
* Active smoking
* Medicated diabetes mellitus (DM)
* Any systemic disease (e.g., wound healing dysfunctions) that could alter the progression of peri-implantitis
* Use of antibiotics and doxycycline, chlorhexidine, and bisphosphonates, within 4 weeks week prior to study participation
* Peri-implant and periodontal treatment within 3 months prior to study participation
* Removable major prosthesis or major orthodontic appliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 6 months
  Change in the inflammatory parameter BOP. A full-mouth assessment at six sites per tooth:
  * Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus
  * Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent"
  * BOP reported as the percentage (%) of sites with positive findings
  * Calculation formula: number of bleeding sites/ 6 times number of teeth

SECONDARY OUTCOMES:
Active matrix metalloproteinase 8 (aMMP-8) | 6 months
  The oral rinse fluid sample collection and the aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
Inflammatory marker total MMP-8 analysis | 6 months
  Measurement of pro and active MMP-8. Units: ng/ml.
Inflammatory marker total MMP-9 analysis | 6 months
  Measurement of pro and active MMP-9. Units: ng/ml.
Inflammatory marker total MMP-2 analysis | 6 months
  Measurement of pro and active MMP-2. Units: ng/ml.
Inflammatory marker total TIMP analysis | 6 months
  Units: ng/ml.
Interleukins analysis | 6 months
  Units: pg/ml.
Total calprotectin analysis | 6 months
  Salivary calprotectin. Units: microgram/ml.
Peridontal Pocket Depth (PPD) | 6 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Visual Plaque Index( VPI) | 6 months
  Assessment of six index teeth, measured at four sites per tooth
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth
Clinical Attachment Level (CAL) | 6 months
  A full-mouth assessment, measured at six sites per tooth
  - Assessed as the distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket (mm)
  The measurements to calculate CAL:
  * distance from the gingival margin to the CEJ and PPD
  * in recession: PPD + gingival margin to the CEJ
  * in tissue overgrowth: PPD - gingival margin to the CEJ
Bacterial flora | 6 Months
  Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis
  - Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Adverse events | 6 months
  Any suspicion of an adverse event related to the investigational device, the treatment method, or the study protocol.
OHIP-14 questionnaire | 6 months
  - Measures people's perception of the social impact of oral disorders on their well-being.
  Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. (Slade GD 1997). Responses are made on a 5-point scale (from 0 = never, to 4 = very often).

OTHER OUTCOMES:
Mobility assessment | 6 months
  Manual assessment of the template movement, mobility testing sideways, and up and down
  - Scoring in numbers 0 - 3
Suppuration index | 6 months
  - Visual assessment of the amount of pus, scoring: 0: No suppuration or exudate present
  1. Minimal suppuration or exudate present
  2. Moderate suppuration or exudate present
  3. Severe suppuration or exudate present

CONTACTS AND LOCATIONS:
Overall Officials: Nilminie Rathnayake, Assoc Prof, Principal Investigator — University of Helsinki
Locations (1):
- Södertandläkarna AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berglundh T, Jepsen S, Stadlinger B, Terheyden H. Peri-implantitis and its prevention. Clin Oral Implants Res. 2019 Feb;30(2):150-155. doi: 10.1111/clr.13401. Epub 2019 Feb 3. PMID 30636066
- [Background] Jepsen S, Berglundh T, Genco R, Aass AM, Demirel K, Derks J, Figuero E, Giovannoli JL, Goldstein M, Lambert F, Ortiz-Vigon A, Polyzois I, Salvi GE, Schwarz F, Serino G, Tomasi C, Zitzmann NU. Primary prevention of peri-implantitis: managing peri-implant mucositis. J Clin Periodontol. 2015 Apr;42 Suppl 16:S152-7. doi: 10.1111/jcpe.12369. PMID 25626479
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Kassebaum NJ, Smith AGC, Bernabe E, Fleming TD, Reynolds AE, Vos T, Murray CJL, Marcenes W; GBD 2015 Oral Health Collaborators. Global, Regional, and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries, and Risk Factors. J Dent Res. 2017 Apr;96(4):380-387. doi: 10.1177/0022034517693566. PMID 28792274
- [Background] Lang NP, Suvan JE, Tonetti MS. Risk factor assessment tools for the prevention of periodontitis progression a systematic review. J Clin Periodontol. 2015 Apr;42 Suppl 16:S59-70. doi: 10.1111/jcpe.12350. PMID 25496279
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- See also: Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019) — https://doi.org/10.1007/s41547-019-00056-9
- See also: Gomes SC, Romagna R, Rossi V, Corvello PC, Melchiors-Angst PD. Supragingival treatment as an aid to reduce subgingival needs: a 450-day investigation Braz. oral res. 28 (1) 2014 — https://doi.org/10.1590/S1806-83242014.50000004
- See also: Levine JI. Medications that increase photosensitivity. FDA document Dec 1990. — https://www.fda.gov/media/75892/download
- See also: Nikinmaa S, Alapulli H, Auvinen P, et al. (2020) Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS ONE 15(5) — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0232775
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. Parkinsonism and Related Disorders 38: 61-67 — https://doi.org/10.1016/j.parkreldis.2017.02.026